CLINICAL TRIAL: NCT05190601
Title: How Valuable is Uroflowmetry in Children With Enuresis Nocturnal?
Brief Title: Uroflowmetry in Children With Enuresis Nocturnal
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Clinical Professor, Hisar Intercontinental Hospital
Other Study IDs: 14.102021/1600
Record Dates: First submitted 2021-12-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Enuresis
Keywords: enuresis nocturna; uroflowmetry; child
MeSH Terms: conditions — Enuresis; Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Group 1: Enuresis nocturna with children
  Interventions: Device: uroflowmetry

INTERVENTIONS:
Device: uroflowmetry — Qmax(ml/s),Qav(ml/s),Volume (ml)

SUMMARY:
Background: Enuresis nocturna is an important social and psychological problem in children. Uroflowmetry is an important test used to investigate lower urinary tract symptoms..

Objective:To evaluate the uroflowmetry (UFM) results of children with nocturnal enuresis (NE).

Method:

The uroflowmetry findings of healthy and visualized children without any urinary symptoms and who were prospectively admitted to the urology and pediatric surgery outpatient clinic with the complaint of Enuresis nocturna between January 2020 and July 2021 were compared. Information (anamnesis, physical examination, radiology results and laboratory tests) and uroflowmetry results of NE and healthy children included in the study were recorded.

DETAILED DESCRIPTION:
SMale and Female,

ELIGIBILITY:
Inclusion Criteria:

Primer monosymptomatic enuresis nocturna

Exclusion Criteria:

Urinary infectious Diabetes Spina bifida, Epispadias, Hipospadias VUR Extrophia Vesica Epilepsy Cerebral Palsy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric,primary monosymptomatic enuresis nocturna, 6-16 years, without comorbidity
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
uroflowmetry | 2 years
  ml/s

CONTACTS AND LOCATIONS:
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)